CLINICAL TRIAL: NCT03285061
Title: Excess Opioid Disposal Following Orthopedic Foot and Ankle Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Christopher Chiodo, Attending Orthopedic Surgeon and Chief of the Foot and Ankle Service at the Brigham and Women's and Faulkner Hospitals, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2017P002031
Record Dates: First submitted 2017-09-14; First posted 2017-09-15 (Actual); Results first posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Medication Disposal; Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard Disposal Instructions (No Intervention): These patients will receive standard instructions on proper disposal of excess pain medication following orthopedic foot and ankle surgery. They will be asked complete a survey at their 6 post operative follow-up on excess medication disposal.
- At Home Disposal (Experimental): With patients' prescription for post operative pain medication, a Deterra portable drug deactivation system will be provided, along with instructions on proper use. They will be asked complete a survey at their 6 post operative follow-up on excess medication disposal.
  Interventions: Device: Deterra Drug Deactivation System

INTERVENTIONS:
Device: Deterra Drug Deactivation System — A portable bag that will neutralize and dissolve excess medication, rendering it completely unusable and safe for landfill disposal. The system meets FDA and DEA standards for at home disposal systems.
  Arms: At Home Disposal

SUMMARY:
This study aims to survey the drug disposal methods of orthopedic foot and ankle patients with excess pain medication following and operation. The study is a randomized control trial comparing the use of FDA approved at home disposal methods to current clinical methods of recommending disposal at medication drop off locations.

ELIGIBILITY:
Inclusion Criteria:

* This study will include foot and ankle orthopedic patients at Brigham and Women's Hospital undergoing a surgical procedure.

Exclusion Criteria:

* Those under age 18 will be excluded from this study, as their variation in care could affect the data. We will also exclude adults with impaired decision-making capacity and adults who take methadone or have a history of prior opioid dependence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Chiodo, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers or organizations.

REFERENCES:
- See also: Deactivation System Website — http://deterrasystem.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Disposal Instructions | At Home Disposal
Started | 37 | 38
Completed | 36 | 36
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Disposal Instructions | At Home Disposal | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 36 | 70
  >=65 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 27 | 51
  Male | 13 | 11 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Safely Disposed The Excess Medication
Description: Patients will be given a survey to obtain their method of disposal for excess post-operative pain medication.
Time Frame: 6 weeks
Population: These two populations constitute a subgroup of all patients initially enrolled in the study.
  Specifically, these two populations constitute those patients that had leftover medications (as opposed to all patients who were enrolled in the trial).
  For this reason, these numbers are disparate from those of the Results Participant Flow.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Disposal Instructions | At Home Disposal
Number analyzed (Participants) | 21 | 26
Participants | 8 | 22

ADVERSE EVENTS:
Time Frame: 6 months
Description: All-Cause Mortality and Serious Adverse Events were not monitored/assessed. This was a survey study with minimal risks. It was anticipated that the questionnaires had no affiliated risk of physical or emotional harm.
Arm/Group | Standard Disposal Instructions | At Home Disposal
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/37 | 0/38

LIMITATIONS AND CAVEATS:
* Single site study: results may not be replicable in other settings or in patients undergoing other procedures
* Potential for reporting bias
* Patients may have felt social pressure to properly dispose of medication
* Since the time of this study, the FDA has conditionally endorsed flushing unused dangerous medications down the toilet in instances in which a take back location is not available.
* Amounts initially prescribed and leftover were not recorded

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT03285061/Prot_001.pdf
  • Statistical Analysis Plan (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT03285061/SAP_003.pdf